CLINICAL TRIAL: NCT07382583
Title: Development of a Shared Decision Tool to Facilitate Uptake of the Levonorgestrel-releasing Intrauterine System for the Primary Prevention of Endometrial Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1540; NCI-2026-00500 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2026-01-22; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Levonorgestrel; Intrauterine Systems; Prevention; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Identify decisional needs, patient values and experiences
  Interventions: Other: Survey using a questionnaire
- Phase 2: Develop and pilot test a web-based shared medical decision tool
  Interventions: Other: Survey using a questionnaire

INTERVENTIONS:
Other: Survey using a questionnaire — Patient Preference Utility Assessment and Questionnaires

SUMMARY:
To develop an educational tool to help patients and healthcare professionals make informed decisions about endometrial cancer and available prevention options for it (such as the use of a levonorgestrel-releasing intrauterine system [LNG-IUS]).

DETAILED DESCRIPTION:
Primary Objectives

The overall goal of this study is to create a personalized decision support educational tool for the use of LNG-IUS as a primary prevention strategy for women at risk of EC. The decision support tool will not replace the consultation with a clinician. Rather, it will help prepare the participant to better understand their options and prepare them for conversations with clinicians when making a decision about use of LNG-IUS. The primary objectives will be accomplished in two phases:

Phase 1 Primary Objective:

1. To identify decisional needs, participant values, and experiences for preferences regarding LNG-IUS through a mixed-methods approach

Phase 2 Primary Objective:

1. To develop and field-test a novel web-based SDM tool in English and Spanish incorporating a personalized EC risk calculator and focused on LNG-IUS as a primary prevention strategy

ELIGIBILITY:
Inclusion Criteria:

1. Unaffected women

   1. Must be at least 18 years old
   2. Must read and speak English or Spanish
   3. Must be premenopausal
   4. Must not have a prior history of EC or complex atypical hyperplasia
   5. Must provide written, informed consent
   6. No physical, psychological, or cognitive impairments that would preclude participation in an interview as determined by the PI or study team member
2. Affected women

   1. Must be at least 18 years old
   2. Must read and speak English or Spanish
   3. Must have a prior history of EC or complex atypical hyperplasia
   4. Must provide written, informed consent
   5. No physical, psychological, or cognitive impairments that would preclude participation in an interview as determined by the PI or study team member
3. Healthcare Providers

   1. Physicians or advanced practice providers (physician assistants, nurse practitioners) from Family Medicine, Obstetrics & Gynecology, Internal Medicine, or Endocrinology
   2. Must be at least 18 years old
   3. Must read and speak English or Spanish
   4. Must provide written, informed consent for qualitative interviews

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2026-07-09 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Patient Utility Questionnaire | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Larissa A Meyer, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The Harris Health System (LBJ), Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org